CLINICAL TRIAL: NCT03910101
Title: Long-term Efficacy of Spasticity-correcting Surgery and Botulinum Toxin Injections for Upper Limb Spasticity Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Theno1RCT
Record Dates: First submitted 2019-03-06; First posted 2019-04-10 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Spasticity, Muscle; Spinal Cord Injuries; Traumatic Brain Injury; Stroke; Upper Extremity Paresis
MeSH Terms: conditions — Muscle Spasticity; Spinal Cord Injuries; Brain Injuries, Traumatic; Stroke; Paresis | interventions — Rehabilitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hand surgery and intensive rehabilitation (Active Comparator): The surgical treatment for reducing spasticity comprises lengthening of tendons, muscle release and occasionally correction of deformities. Lengthening of a tendon or releasing a muscle from its insertion, results in relaxation of the whole muscle-tendon unit. Hence, the spasticity is not gone, but reduced in strength.
  The tendon lengthening procedures is performed by a stair-step incision technique followed by reattachment in the lengthened position using a side-to-side, cross-stich technique. The load to failure of the sutured tendon is approximately 200Newton, which gives a sufficient safety margin for early active mobilization of the tendons involved. This suture technique thus enables active training directly after surgery.
  Postoperative rehabilitation includes wrapping and a custom-made splint, for day and night use, muscle activation and passive stretching 2-4 times per day without the splint.
  Interventions: Procedure: Hand surgery and intensive rehabilitation
- Botulinum toxin injections (Active Comparator): Botulinum toxin injections are given in spastic muscles of the upper extremity. Dosage and number of injections per muscle vary depending on the degree and extent of spasticity. For optimal effect on hand function, botulinum toxin is accompanied by the treatment of individualized exercise and splinting when needed.
  Interventions: Procedure: Hand surgery and intensive rehabilitation

INTERVENTIONS:
Procedure: Hand surgery and intensive rehabilitation — Spasticity-correcting upper-limb surgery comprised lengthening of tendons, release of muscles, and occasionally correction of deformities. Rehabilitation starts the first post-operative day and comprised physiotherapy and occupational therapy. Patients are also taught a home-training program. Up to 1 week of intensive in-hospital rehabilitation followed 3 weeks after surgery and a new home-training program are designed.
  Other Names: Botulinum toxin injections and rehabilitation

SUMMARY:
Spasticity - a variety of motor over-activity and part of the upper motor neuron syndrome - is a common cause of impaired motor function after brain injuries of different etiologies. In addition, it may cause pain and impaired hygiene, contractures, deformities etc. Spasticity has been reported in 30 to 90% of patients with stroke, traumatic brain injury (TBI), incomplete spinal cord injury (SCI) and cerebral palsy (CP).

Spasticity therapy has emerged as an important approach to alleviate related symptoms. Positive effects on spasticity are well recognized following systemic and intra-thecal pharmacological treatment, as well as after intra-muscularly injected substances; the effect of the latter is, however, of limited duration. While pharmacological spasticity therapy has been applied for decades, surgical procedures remain fairly uncommon in adults with spasticity, but not in pediatric patients with CP, and outcomes after surgical treatment are scarcely described in the literature.

The study center is a specialized unit initially focused on reconstructive as well as spasticity reducing surgery in the upper extremities for SCI patients. Subsequently, patients with spasticity also due to various other Central nervous system diseases have been referred to the center for surgical treatment. Studies describing the effect of spasticity-reducing surgery in the upper extremities are rare and the group is heterogeneous. The aim of the study is evaluating the long-term efficacy of spasticity-correcting surgery versus BoNT in patients with disabling UL spasticity. As a secondary aim, we want to compare the peak effects of the two treatments, Botulinum toxin injections and spasticity-correcting surgery.

DETAILED DESCRIPTION:
Study design and participants This study used a pretest-posttest quasi-experimental design.

Study participants are recruited using two parallel procedures. I) Review of a hospital-based register of patients who had been treated or referred to the tonus clinic identified eligible patients, who were then sent information about the study, along with their contact information to the researcher responsible for the study. II) Patients with ongoing BoNT treatment who had been referred to the Center for Advanced Reconstruction of Extremities (C.A.R.E.), and were eligible for the present study were informed about the study and enrolment procedure.

All presumptive study participants will undergo a screening procedure by the primary examiner, to assess whether they met the study's eligibility criteria. Written informed consent will be obtained if the patient met the inclusion criteria and consented to participate. All patients are offered either of the two treatment methods, the treatment allocation are based on individual preferences. The study will be conducted in accordance with relevant ethical guidelines (Declaration of Helsinki).

The primary outcome measure are muscle tone, measured using the Modified Ashworth Scale (MAS). The single-item MAS was measured on a six-point scale from 0 (no increase in muscle tone) to 4 (affected part rigid in flexion or extension), with an additional point allocated at 1+ (slight increase in muscle tone). As such, the MAS provides a single score to represent spasticity in a specific movement. For analysis, the MAS scores of the treated muscles were summed to obtain a "composite spasticity score" for each participant.

Secondary outcomes includes measures within, body function, activity and Participation.

The calculation of sample size was based on the a priori defined difference to be detected, with an alpha level of 5% and a power goal of 80%, as well as the primary outcome variable MAS and previous findings. Provide a number of 14 participants in each of the two groups. We expected a dropout rate of 15%, and therefore aimed to include 17 individuals in each group to achieve 80% power.

Between-group differences and within-group differences in treatment efficacy will be analysed by comparing pretest-posttest changes.

ELIGIBILITY:
The eligibility criteria for this study were as follows: 1. 18 years or above; 2. Problematic spasticity, characterised by a velocity-dependent increase in tonic stretch reflexes or intermittent or sustained involuntary muscle activity in the UL after stroke, TBI, or SCI; and 3. Patients treated at least 6 months after the injury event; and 4. Ongoing BoNT treatment in the UL, 5. A minimum of 3 months passed since the last BoNT injection: 6. At least two muscles in the hand and wrist were considered for treatment 7. For the BoNT group, a community occupational or physical therapist was assigned for post BoNT treatment; 8. For the surgery group, medically stable to undergo surgery; 9. No other severe UL injuries affecting the functional level.

Exclusion Criteria:

* Under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Change is being assessed with Modified Ashworth Scale | Change from baseline and at the the time points 4-6weeks and 6months
  0-5 scale that quantify the degree of resistance to passive movement of the target muscle group

SECONDARY OUTCOMES:
Change is being assessed with Visual Analog scale (VAS) | Change from baseline and at the the time points 4-6weeks and 6months
  for pain, patient's self-rating of general arm-hand function (usefulness), appearance of the hand and self-rating spasticity. Visual Analog Scale is a straight horizontal line of fixed length, 100 mm. The ends are defined as the extreme limits of the parameter to be measured. Orientated from the left no; pain, spasticity, problem with appearance to the right worst possible; pain, spasticity, problem with appearance. In the general hand function question the scale goes from left side no hand function to the right side best possible hand function. In the pain, spasticity and appearance question a high number indicate a worse outcome, in the general hand function question a high number represent a better outcome. Respondents specify their level of agreement to the statement by indicating a position along the line.
Change is being assessed with goniometry | Change from baseline and at the the time points 4-6weeks and 6months
  to measure joint resting position and passive and active range of motion (ROM). Higher numbers indicates better outcomes
Change is being assessed with Jamar dynamometer | Change from baseline and at the the time points 4-6weeks and 6months
  grip strength, higher scores indicates better outcomes
Change is being assessed with pinch gauge | Change from baseline and at the the time points 4-6weeks and 6months
  measuring strength in the two- point tip- and lateral key-pinch, Higher scores indicates better outcomes
Change is being assessed with opening of the hand passive, Active and resting position | Change from baseline and at the the time points 4-6weeks and 6months
  Five step scale that goes from closed, 1/4 opened, 1/2 opened, 3/4 opened, open hand. Higher scores indicates better outcomes.
Change is being assessed with The Canadian Occupational Performance Measure (COPM) | Change from baseline and at the the time points 4-6weeks and 6months
  measuring performance and satisfaction of therapy regarding the most important activity limitations due to spasticity (up to 5) as chosen and assessed by the patient on a scale from 1-10, higher number indicates better outcomes.
Change is being assessed with Grasp and Release Test (GRT) | Change from baseline and at the the time points 4-6weeks and 6months
  assessing the patients' ability to grasp, move, and release 6 objects of varying weight and size during 30 seconds. Higher scores indicates better outcomes.
Change is being assessed with Arm Activity Measure (ArmA) | Change from baseline and at the the time points 4-6weeks and 6months
  a patient reported outcome measure of active and passive function in the hemiparetic upper limb. Lower scores indicates better outcomes.
Change is being assessed with Cylinder test | Change from baseline and at the the time points 4-6weeks and 6months
  the test is measuring the opening and grasp ability of the patient's hand. The test evaluate four different way of grasping; normal one hand grip, adapted one hand grip, two hand grip and adapted two hand grip. The test consists cylinders in 15 different sizes from 10mm to 150mm. The cylinder test enables measuring progress of opening the hand during rehabilitation or before and after surgery. Higher scores indicates better outcomes.
Change is being assessed with Functional score | Change from baseline and at the the time points 4-6weeks and 6months
  Grade the upper limb function (1-4). Description
  1. Absence of useful active mobility and uneasy and painful passive mobilization, making difficult to dress and wash
  2. Easy passive mobilization but without any useful voluntary movements
  3. Slight but useful voluntary motor function
  4. Good active mobility with the possibility of prehension in the hand and fingers. Higher numbers indicates better outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Lina Bunketorp Kall, PhD, Study Chair — University of Gothenburg, Sahlgrenska academy
Locations (1):
- Sahlgrenska University Hospital, centrum for advanced reconstruction of extremities, Mölndal, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No